CLINICAL TRIAL: NCT00910052
Title: Routine Use of Fibrin Sealant Does Not Reduce Postoperative Wound Complications in Patients Undergoing Renal Transplantation: A Randomized Controlled Trial
Brief Title: Fibrin Sealant in Renal Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin County Medical Center, Minneapolis (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20032206
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Renal Transplantation
Keywords: randomised; controlled; double blinded

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrin sealant (Experimental): received intraoperative fibrin sealant
  Interventions: Device: Tisseelä fibrin sealant
- Control (No Intervention): No fibrin sealant

INTERVENTIONS:
Device: Tisseelä fibrin sealant — Fibrin sealant applied intraoperatively
  Arms: Fibrin sealant

SUMMARY:
Background: Post-operative wound complications arise in as many as 50% of kidney transplant recipients. Fibrin sealants have been used in many areas of surgery in attempt to reduce the accumulation of post-operative fluid collections with varying success. The use of fibrin products has been proposed as a means of reducing local wound complications in the immunocompromised renal transplant recipient but as yet has not been studied.

Methods: 145 patients were enrolled and 141 patients were randomized (74 Tisseelä fibrin sealant, 67 No Tisseelä fibrin sealant) in a prospective manner to receive fibrin sealant or not at the time of their renal transplant. Patients were analyzed per the randomization assignment. The operating team was blinded to the decision until after the iliac fossa dissection was complete. The sealant was applied via aerosol to the iliac fossa and renal allograft hilum after completion of the neoureterocystostomy in 5 ml quantity. Clinical and radiographic data were reviewed through the usual 8-week follow-up transplant ultrasound. Patients in whom the peritoneum was entered were excluded from data analysis. The incidence of lymphocele, wound infection, dehiscence, clinically significant hematoma as defined by necessitating incision and drainage, and urine leak was recorded.

ELIGIBILITY:
Inclusion Criteria:

* All renal transplant recipients

Exclusion Criteria:

* Patients declining study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2003-05; Primary Completion 2006-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
presence of postoperative fluid collection

SECONDARY OUTCOMES:
wound infection
wound dehiscence

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States